CLINICAL TRIAL: NCT03879681
Title: SNAKES UK: a Pilot Trial of Jelly Snakes to Prevent Postoperative Nausea and Vomiting in Kids After ENT Surgery
Brief Title: SNAKES Trial: Jelly Snakes to Prevent PONV in Kids After ENT Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Thomas Engelhardt (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Thomas Engelhardt, Consultant, National Health Service, United Kingdom
Organization: National Health Service, United Kingdom (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Snakes UK
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: POSTOP NAUSEA VOMITING; Tonsillectomy; Adenoidectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention)
- Jelly Snakes (Experimental)
  Interventions: Dietary Supplement: Jelly confectionary Snakes

INTERVENTIONS:
Dietary Supplement: Jelly confectionary Snakes — The participants will be randomized by computer generated randomisation to receive either the jelly snake (n=120) or no intervention (n=120) apart from standard institutional management.
  All children randomised into the snake group will be offered a chewy jelly snake once alert and cooperative in PACU or on the ward once University of Michigan Sedation Scale (UMSS) is 025,26. The UMSS is a simple observational tool that assesses the level of alertness on a five-point scale ranging from 1 (wide awake) to 5 (unarousable with deep stimulation).
  The children randomized into the control group will receive a chewy jelly snake as a treat at discharge.
  Arms: Jelly Snakes

SUMMARY:
Postoperative nausea and vomiting in children is a common phenomenon, particularly after ear nose and throat (ENT) surgery. While it affects up to 80% of patients who do not receive preventative medication during their operation, more than 1 in 5 children still suffer from postoperative nausea and vomiting after tonsillectomy even when given 2 medications to prevent it. Nausea and vomiting after an operation (postoperatively) particularly following tonsillectomy can be very painful and distressing for the child and their carer. Vomiting may also increase the risk of postoperative bleeding, a serious complication after the surgery. Postoperative nausea and vomiting is not only one of the main reasons for prolonged hospital stay or re-admission in children; it is also one of the main reasons for dissatisfaction with anaesthesia in children and their families. In adults, a pilot study has found that chewing gum postoperatively can significantly reduce postoperative nausea and vomiting. Chewing and swallowing, results in increased activity in the gut and lessens the effects of medications given under anaesthesia that tend to slow the gut.

However, for young children particularly following anaesthesia, chewing gum may not be a safe option. Therefore, in this pilot study the investigators will investigate if chewing a large jelly confectionary snake after the anaesthetic will help to reduce nausea and vomiting. The children who are enrolled in the study will be randomised to receive a jelly snake or no jelly snake to chew once awake after the surgery. There will be no other changes to the standard management which will be in accordance to institutional guidelines. The investigators will then compare the rates of vomiting between the children who did and did not receive a jelly snake to chew. We will also monitor other oral and food intake and requirements for painkillers, as well as for other potential problems (e.g. delayed discharge) after surgery.

The advantage of using a jelly snake is that it is a simple, inexpensive, non-drug treatment. Parents are very keen to avoid the use of drugs for their children and so would be open to the use of this new approach. For children the jelly snake offers something familiar and an enjoyable solution to their discomfort. The use of jelly snakes could also be a simple intervention that parents could do at home following day case surgery for other procedures. While the jelly snakes are high in sugar, they are comparable to the sugar content of a glass of fruit juice, flavoured milk or soft drinks. Generally, in the investigators' experience, the willingness of parents to allow their children to receive treats in the postoperative period is very high, particularly since all children have a significant time of fasting (at least 6 hours, often longer) for solid foods prior to surgery.

DETAILED DESCRIPTION:
Primary Hypothesis Chewing large jelly snakes will significantly reduce the development of postoperative vomiting in paediatric patients in the first 6 hours after volatile anaesthetic-based general anaesthesia for tonsillectomies +/- adenoidectomies.

Secondary Hypotheses:

1. Jelly snakes will reduce the incidence of nausea in the first 6 hours after tonsillectomy +/- adenoidectomy surgery
2. Jelly snakes will reduce rescue treatments for PONV in the first 6 hours
3. Jelly snakes will reduce the incidence of PONV in the first 24 hours or up until discharge in case of tonsillectomies (whatever occurs first)
4. Jelly snakes will reduce rescue treatments for PONV in the first 24 hours or up until discharge in case of tonsillectomies (whatever occurs first)

Safety Hypotheses:

Children will be able to chew and swallow jelly snakes post-surgery. No jelly snake or parts thereof will be inhaled in those receiving treatment.

Aims This pilot study aims to investigate if chewing jelly confectionary snakes after tonsillectomies +/- adenoidectomies will significantly reduce the incidence of postoperative nausea/vomiting (PONV) in children.

Study Design One site pilot trial of the effectiveness of chewy jelly snakes in the prevention of POV involving the Royal Aberdeen Children Hospital, UK.

ELIGIBILITY:
Inclusion Criteria:

* Volatile anaesthetic-based general anaesthesia
* Written informed parental consent
* Elective tonsillectomy +/- adenoidectomy (+/- myringotomy, EUA ear, grommets or cautery of inferior turbinates')

Exclusion Criteria:

* Plan to use muscle relaxant
* Plan to use topical lignocaine on the vocal cords intraoperatively
* Contraindication to chewy jelly snakes or any of their components e.g. known allergy to any of the ingredients of the chewy jelly snakes or impaired pharyngeal/oesophageal function (e.g. bulbar palsy, achalasia), children with diabetes and vegetarian children
* Contraindication to any protocolised anti-emetic drug (prophylaxis, intervention or rescue)
* Parents/guardians or children who, in the opinion of the investigator, may be unable to understand or give informed consent will be excluded from the study.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative vomiting in paediatric patients in the first 6 hours after volatile anaesthetic-based general anaesthesia for adenoidectomies and / or tonsillectomies | up to 6 hours after the end of the surgery

SECONDARY OUTCOMES:
Incidence of nausea in the first 6 hours post tonsillectomy +/- adenoidectomy surgery in children over 8 years | up to 6 hours after the surgery
• Number of rescue treatments for PONV in the first 6 hours | up to 6 hours after the surgery
• Incidence of PONV in the first 24 hours or up until discharge (whatever occurs first) | Up to 24 hours
• Time to first vomit if applicable (measured from arrival in PACU) | Up to 24 hours
• Time to first meal | Up to 24 hours
• Duration of hospital stay | Up to 48 hours

IPD SHARING:
Plan to Share IPD: Undecided